CLINICAL TRIAL: NCT00122356
Title: Maintaining Skeletal Health in Postmenopausal Women With Surgically Resected Stage I-IIIa Hormone-receptor Positive Breast Cancer Who Are Receiving Anastrozole, Through the Use of Alendronate as Determined by the Osteoporosis Australia Bone Maintenance Algorithm
Brief Title: Bisphosphonate and Anastrozole Trial - Bone Maintenance Algorithm Assessment
Acronym: BATMAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Barwon Health (Other Government)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ALCC 04.02
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Alendronate

ARMS (1):
- Anastrozole and alendronate (Other): Patients will receive anastrozole for 5 years and alendronate for 3 years or anastrozole and alendronate treatment for 5 years.
  Interventions: Drug: Alendronate sodium

INTERVENTIONS:
Drug: Alendronate sodium — 70mg tablets, once weekly
  Other Names: Fosamax; Alendro; Adronat

SUMMARY:
The purpose of this study is to evaluate the use of an oral bisphosphonate (alendronate) in preventing bone loss in postmenopausal women with early breast cancer who are receiving anastrozole therapy, and to determine how long alendronate treatment is needed.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* Adequately diagnosed and treated Stage I-IIIa early breast cancer
* Oestrogen receptor and/or progesterone receptor positive breast cancer
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Hormone replacement therapy (HRT) must be discontinued at least 2 weeks prior to registration
* Any prior tamoxifen taken for a total of 8 weeks or less
* Any prior anastrozole taken for a total of 4 weeks or less
* Anastrozole is clinically indicated to be the best adjuvant strategy
* Signed written informed consent

Exclusion Criteria:

* Clinical or radiological evidence of distant spread of disease
* Prior treatment with bisphosphonates within the past 12 months
* Prior treatment with continuous systemic corticosteroids within the past 12 months
* Prior use of parathyroid hormone for more than 1 week
* Prior use of systemic sodium fluoride for > 3 months during the past 2 years
* Currently treated with any drugs known to affect the skeleton
* Abnormal renal function (serum creatinine greater than or equal to 265.2 mmol/L)
* History of diseases with influence on bone metabolism. Patients with lactose intolerance are also excluded
* Delayed oesophageal emptying such as stricture or achalasia
* Hypersensitivity to alendronate or anastrozole
* Previous or concomitant malignancy within the past 5 years EXCEPT adequately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix
* AST/SGOT and/or ALT/SGPT > 3 x ULN in combination with other laboratory and clinical abnormalities indicating liver insufficiency
* Fracture due to minimal trauma, demonstrated radiologically

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2005-09; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Changes in lumbar vertebra and femoral neck bone mineral density (BMD) T-score after 5 years of anastrozole treatment | 5 years

SECONDARY OUTCOMES:
Percent change in the lumbar vertebra (L2 to L4) and femoral neck BMD | 12 monthly intervals
Biochemical markers of bone turnover (N-telopeptide and bone-specific alkaline phosphatase) and BMD | 6 months after registration and/or 6 months after commencing alendronate
Evaluate the Osteoporosis Australia strategy for bone protection for this patient group | 5 years
Evaluate the clinical fracture incidence cumulative over 5 years | 5 years
Perform an economic analysis of the cost of monitoring and intervention | 5 years
Evaluate the time to disease recurrence/relapse in women treated with anastrozole as adjuvant therapy | 5 years
Evaluate the effects of anastrozole on serum lipid parameters following 6 months therapy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen White, Principal Investigator — Barwon Health
Locations (8):
- Australia (8):
  - Sydney South West Area Health Service, Sydney, New South Wales
  - Tweed Hospital, Tweed Heads, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Maroondah Breast Clinic, East Ringwood, Victoria
  - St Vincent's Health, Fitzroy, Victoria
  - Barwon Health, Geelong, Victoria
  - St John of God Healthcare, Geelong, Victoria
  - South West Healthcare, Warrnambool, Victoria

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716